CLINICAL TRIAL: NCT05592782
Title: Virtual Reality Mindfulness Study
Brief Title: VR Mindfulness Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left UCLA
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB#22-001517
Record Dates: First submitted 2022-10-14; First posted 2022-10-25 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Anxiety; Depression; Stress; Pain, Acute; Pain, Chronic
Keywords: Virtual Reality; Anxiety; Depression; Pain; Mood; Mindfulness; Meditation
MeSH Terms: conditions — Anxiety Disorders; Depression; Acute Pain; Chronic Pain; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Arm (Experimental)
  Interventions: Behavioral: Virtual Reality Based Mindfulness meditation

INTERVENTIONS:
Behavioral: Virtual Reality Based Mindfulness meditation — Participants will undergo a guided VR meditation using a commercial VR application. The meditation will last approximately 15 minutes. Prior to starting and on upon completion of each VR meditation session, participants' state pain, anxiety, depression, and stress will be assessed. For each participant enrolled, baseline and monthly assessments using the DASS-21 and PPI-SFI3a will be performed for three consecutive months.

SUMMARY:
This is an exploratory study investigating the use of virtual reality-based guided mindfulness meditation in improving pain, stress, and mood within various clinical populations. The feasibility of utilizing VR applications within the populations of patients with various specific disease types and clinical settings is a burgeoning area of research. The goal is to establish an association between the use of VR-based mindfulness meditation, and pain, stress, and mood scores.

DETAILED DESCRIPTION:
This is a two-center, multi-site exploratory study conducted within the University of California, Los Angeles Health and Greater Los Angeles VA systems. A total of 60 subjects will be recruited. Screening data will be reviewed to determine subject eligibility. Subjects who meet all inclusion criteria and none of the exclusion criteria will be entered into the study.

Subjects will undergo assessments of stress, depression, anxiety, and pain at baseline, pre- and post-VR guided mediation, and monthly for three months. Each subject can undergo VR-guided meditation session no more than one time per day. In subjects who are hospitalized, an attempt will be made to have the subjects undergo the VR meditation and complete the pre- and post- meditation assessments daily until hospital discharge.

Duration of the study is expected to be 1 year. Each session is expected to last approximately 15 minutes.

Subjects will be given instructions on proper use of the VR devices and how to start the guided meditation software. Once familiar with the device, participants will undergo a guided VR meditation using a commercial VR application. The meditation will last approximately 15 minutes. Prior to starting and on upon completion of each VR meditation session, participants' state pain, anxiety, depression, and stress will be assessed. For each participant enrolled, baseline and monthly assessments using the DASS-21 and PPI-SFI3a will be performed for three consecutive months

ELIGIBILITY:
Inclusion Criteria:

* Adults at least 18 years old
* Able to read and understand English (Guided meditation software has not yet been translated to languages other than English)

Exclusion Criteria:

* Age <18 years old
* Unable to speak, read or understand English language
* Blindness or severe hearing impairment
* Any disability or neurological deficit that would impair subject from using the virtual reality console
* Significant movement disorder
* Vertigo and/or motion sickness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Completion of VR Mindfulness Meditation Session | 2 hours
  Proportion of subjects able to complete VR meditation sessions
State Anxiety | 2 hours
  Change in STAI-6 scores pre- and post-use of VR meditation application
Pain severity | 2 hours
  Change in VAS-100 scores pre- and post-use of VR meditation application

SECONDARY OUTCOMES:
Ease of use and acceptability | 2 hours
  Modified User Satisfaction Evaluation Questionnaire scores after each session
Depression | 2 hours
  Change in BDI-SF scores pre and post-use of VR meditation
Stress | 2 hours
  Change in SSSQ scores pre- and post-use of VR meditation
Long term change in Stress, Anxiety, and Depression | 3 months
  Change in DASS-21 scores monthly for 3 months
Long term change in Pain severity | 3 months
  Change in PROMIS Pain Intensity- Short Form 3a scores over 3 months
Hospital Length of Stay | 4 months
  Compare subject length of stay in hospital to average length of stay for admission diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Arash Naiem, MD, PhD, Principal Investigator — University of California, Los Angeles